CLINICAL TRIAL: NCT03915522
Title: Adductor Canal Block in an Enhanced Recovery Program After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Responsible Party: Principal Investigator, Reis Drudis, Principal Investigator, Institut de Recerca Biomèdica de Lleida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIC-1806
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Total Knee Arthroplasty; Knee Osteoarthritis
Keywords: total kee arthroplasty; adductor canal block; multimodal analgesia
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A simple randomization is made to distribute the included patients in two groups: Standard Group and Intervention Group. A table of random numbers is used, first selecting the starting point and later the movement direction remains constant throughout the whole table. The even numbers are allocated in the standard group and the odd ones in the intervention group.
Who Masked: Participant, Outcomes Assessor
Masking Description: All patients included in the study are transferred the day after the total knee arthroplasty surgery to the postoperative resuscitation unit.
  A sterile dressing of the lower extremity is performed and after the adductor canal is identified with ultrasound image, a medial leg puncture is done with or without doing the canal adductor block. At the end all patients have a sterile apposite on the puncture site.
  All variables and outcomes are collected and registered by people not involved in the realization of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor Canal Block (Experimental): Patients will receive multi-modal analgesia (oral, intravenous and local infiltration anesthesia) for pain management following total knee arthroplasty and in the first postoperative day a single adductor canal block wiht 20cc of 0.5% Ropivacaine using ultrasound guidance .
  Interventions: Procedure: Single adductor canal block
- Placebo Comparator (Placebo Comparator): Patients will receive multi-modal analgesia (oral, intravenous and local infiltration anesthesia) for pain management following total knee arthroplasty and in the first postoperative day a sham adductor canal block with 2ml of 1% subcutaneous lidocaine at the level of the adductor canal using ultrasound guidance.
  Interventions: Procedure: Simulated adductor canal block

INTERVENTIONS:
Procedure: Single adductor canal block — The operated leg is slightly externally rotated and prepared for a block with 2% chlorhexidine and sterile dressing. The adductor canal is identified using ultrasound image at the mid-thigh level and after a subcutaneous injection of 2 ml of 1% lidocaine a total of 20 ml of 0'5% ropivacaine is injected into the canal using a 22 gauge ultrasound-visible needle. In the end, a sterile apposite is placed at the puncture site
  Arms: Adductor Canal Block
Procedure: Simulated adductor canal block — The operated leg is slightly externally rotated and prepared with 2% chlorhexidine and sterile dressing. The adductor canal is identified using ultrasound image at the mid-thigh level and at this leve a subcutaneous injection of 2 ml of 1% lidocaine . After, a sterile apposite is placed at the puncture site.
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to assess the effectivity of adductor canal block performed the day after total knee arthroplasty surgery in reducing pain and improving walking ambulation ability and muscle strength.

DETAILED DESCRIPTION:
Overview: total knee arthroplasty is a painful procedure. According to our institutional pain registers the worst pain appears in postoperative day one, which could be related to the use of effective but short analgesic intraoperative techniques like periarticular local analgesic infiltration and intravenous multimodal analgesia.

The aim: to asses if adductor canal block performed the day after primary total knee arthroplasty (16-20 hours postoperative) improves analgesia without motor blockade and impairment of early ambulation ability.

Primary Hypothesis: adductor canal block performed 16-20 hours after primary total knee arthroplasty improves postoperative analgesia.

Secondary Hypothesis: adductor canal block performed 16-20 hours after primary total knee arthroplasty improves ability of early ambulation, adductor and quadriceps strength after primary total knee arthroplasty.

The objectives:

1. To compare postoperative pain control effects between adductor canal block and placebo block.
2. To assess the improvement of ability of early ambulation and extent of motor blockade after primary total knee joint replacement surgery between the groups of patients.
3. To estimate variations in quadriceps and adductor muscle strength in the two groups of patients.
4. To asses related side effects to adductor canal nerve block.
5. To asses variations in length of stay between the two groups.

Methods:

The prospective, double-blinded study includes American Society of Anesthesiologists (ASA) physical status I-III in preoperative assessment, aged 18-85 years, admitted for primary total knee arthroplasty. Preoperatively a simple randomization is made to distribute the included patients in two groups: Standard Group and Intervention Group. A table of random numbers is used, first selecting the starting point and later the movement direction remains constant throughout the whole table. The even numbers are allocated in the Standard Group and the odd ones in the Intervention group. The anesthesiologist performing the block will be aware of the treatment, but the participant subject and outcomes assessor will be blinded to the group assignment.

During the perioperative period all patients from both groups will receive a standardized anesthetic and analgesic treatment: premedication with midazolam 2.5-5 mg and dexamethasone 0'1 mg/kg, spinal anesthesia with 10mg of hyperbaric bupivacaine and intravenous propofol during the surgery for sedation. As analgesia paracetamol 1gr plus dexketoprofen 50 mg. The local infiltration analgesia will be performed in a protocolized manner during the surgery with ropivacaine 0'2% 120 cc mixed with 0'6 mg adrenaline and at the end of surgery with ropivacaine 0'2% 40cc for subcutaneous infiltration. Two doses of 0'1mg/kg tranexamic acid are administrated unless contraindication, first one 30 min before skin incision and second one three hours later.

Postoperative analgesia will be administrated to both groups of patients with ibuprofen 600 mg/8h and paracetamol 1gr/6h. Opioids will be available to patients as intravenous boluses of tramadol 1mg/kg if pain numerical rate score (NRS) > 3 at rest or > 5 at movement.

All patients included in the study are transferred to post-anesthesia reanimation unit 16-20h after surgery, in postoperative day one. The operated extremity is slightly externally rotated and prepared for the block with 2% chlorhexidine and sterile dressing and the adductor canal is identified with ultrasound image at the mid-thigh level. In standard group patients a sham adductor canal block with 2ml of 1% subcutaneous lidocaine is done. In intervention group patients an adductor canal block with a 22 Gauge ultrasound-visible needle and 20 ml of 0'5% ropivacaine is done. At the end all patients have a sterile apposite on the puncture site.

Postoperative pain will be assessed 15 minutes before the procedure (adductor or sham block), 2 hour, 24 hour post and also in the three nursing rounds (morning, afternoon, night) the first 72 hours after surgery. The pain numeric rating scale (NRS) is used (from 0 - no pain to 10 - worst imaginable pain) at rest and during active knee flexion. The requirement of additional opioids and their side effects (if any) will be recorded.

Knee extensor and adductor muscle strength is measured using a hand-held dynamometer (Baseline Digital Hydraulic Push Pull Dynamometer R)) immediately prior to surgery, in first postoperative, day immediately before the procedure, 2 hours and 24 hour postprocedure.

Patients ability of early ambulation is evaluated using ten meter walk test (TMWT) in the first and second postoperative day every 12h.

The success rate of the block is assessed by testing for sensation of cold and pinprick stimulus at the medial midcalf using a 3-point scale (2 = normal sensation, 1 = decreased sensation, 0 = no sensation) 2 hours after block.

The length of hospital stay and rate of complications (if any), will be recorded in both groups of patients. Complications will be graded as local complications (hematoma, wound complications…), block complications (falls, vascular injection…), urinary complications (acute urine retention, renal failure…) and general complications (neurological, respiratory, cardiological…).

According to study protocol, both groups of patients will be compared in terms of postoperative pain control, opioid consumption, postoperative nausea and vomiting, quadriceps strength, adductor strength, ability of early ambulation, length of hospitalization and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective unilateral total knee arthroplasty
* American Society of Anesthesiologist (ASA) class 1-3
* Adults aged 18-85 years old

Exclusion Criteria:

* Contraindications of the adductor canal block.
* Contraindications of the local infiltration analgesia technique.
* Chronic kidney disease
* Surgery to be performed under general anesthesia.
* Opioid treatment > 30 mgr morphine or equivalent for more than 3 months time.
* Neuropathic ipsilateral pain.
* Inability to understand study procedures.
* Not acceptance of the procedure (adductor canal block or local infiltration analgesia).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-09-02 (Estimated); Study Completion 2019-09-02 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative pain score at rest and knee flexion: Numerical Rating Scale | Registered immediately prior to surgery, first postoperative day immediately prior to procedure, 2 hours postprocedure and every 8 hours the first three days in the orthopedic ward.
  Assessed using a Numerical Rating Scale (NRS) from 0 to 10

SECONDARY OUTCOMES:
Knee extensor muscle strength | Immediately prior to surgery, first postoperative day immediately before the intervention , 2 and 24 hours postintervention
  Measured using a hand-held dynamometer
Adductor muscle strength | Immediately prior to surgery, first postoperative day immediately before the intervention , 2 and 24 hours postintervention
  Measured using a hand-held dynamometer
Ability to walk with ten meter walk test | First and second postoperative day every 12 hours
  Measured with the ten meter walk test (TMWT)
Rate of pain rescue treatments. | First 72 hours following surgery
  Rate of intravenous opioid needed by the patients.
Rate of opioid side effects. | First 72 hours following surgery
  Rate of episodes of dizziness or nausea or vomit after opioid intake.
Length of hospital stay | From date to operation until the data of discharge home, assessed up to 1 month
Rate of adductor canal block complications | First 72 hours following surgery
  Including: local swelling, hematoma, vascular or neurological lesion and falls.
Rate of surgery local complications | From date to operation until the data of discharge home, assessed up to 1 month
  Including, hematoma, wound infection, arthroplasty infection, vascular or neurological lesion.
Rate of medical complications | From date to operation until the data of discharge home, assessed up to 1 month
  Including neurological, cardiological, urological and respiratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitary Santa Maria, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Andersen LO, Kehlet H. Analgesic efficacy of local infiltration analgesia in hip and knee arthroplasty: a systematic review. Br J Anaesth. 2014 Sep;113(3):360-74. doi: 10.1093/bja/aeu155. Epub 2014 Jun 17. PMID 24939863
- [Background] Xu CP, Li X, Wang ZZ, Song JQ, Yu B. Efficacy and safety of single-dose local infiltration of analgesia in total knee arthroplasty: a meta-analysis of randomized controlled trials. Knee. 2014 Jun;21(3):636-46. doi: 10.1016/j.knee.2014.02.024. Epub 2014 Mar 13. PMID 24704172
- [Background] Sawhney M, Mehdian H, Kashin B, Ip G, Bent M, Choy J, McPherson M, Bowry R. Pain After Unilateral Total Knee Arthroplasty: A Prospective Randomized Controlled Trial Examining the Analgesic Effectiveness of a Combined Adductor Canal Peripheral Nerve Block with Periarticular Infiltration Versus Adductor Canal Nerve Block Alone Versus Periarticular Infiltration Alone. Anesth Analg. 2016 Jun;122(6):2040-6. doi: 10.1213/ANE.0000000000001210. PMID 27028771
- [Background] Fajardo M, Collins J, Landa J, Adler E, Meere P, Di Cesare PE. Effect of a perioperative intra-articular injection on pain control and early range of motion following bilateral TKA. Orthopedics. 2011 May 18;34(5):354. doi: 10.3928/01477447-20110317-11. PMID 21598890
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Jaeger P, Grevstad U, Henningsen MH, Gottschau B, Mathiesen O, Dahl JB. Effect of adductor-canal-blockade on established, severe post-operative pain after total knee arthroplasty: a randomised study. Acta Anaesthesiol Scand. 2012 Sep;56(8):1013-9. doi: 10.1111/j.1399-6576.2012.02737.x. Epub 2012 Jul 26. PMID 22834681
- [Background] Andersen HL, Gyrn J, Moller L, Christensen B, Zaric D. Continuous saphenous nerve block as supplement to single-dose local infiltration analgesia for postoperative pain management after total knee arthroplasty. Reg Anesth Pain Med. 2013 Mar-Apr;38(2):106-11. doi: 10.1097/AAP.0b013e31827900a9. PMID 23222363
- [Background] Jaeger P, Koscielniak-Nielsen ZJ, Schroder HM, Mathiesen O, Henningsen MH, Lund J, Jenstrup MT, Dahl JB. Adductor canal block for postoperative pain treatment after revision knee arthroplasty: a blinded, randomized, placebo-controlled study. PLoS One. 2014 Nov 11;9(11):e111951. doi: 10.1371/journal.pone.0111951. eCollection 2014. PMID 25386752
- [Background] Hanson NA, Allen CJ, Hostetter LS, Nagy R, Derby RE, Slee AE, Arslan A, Auyong DB. Continuous ultrasound-guided adductor canal block for total knee arthroplasty: a randomized, double-blind trial. Anesth Analg. 2014 Jun;118(6):1370-7. doi: 10.1213/ANE.0000000000000197. PMID 24842182
- [Background] Kuang MJ, Xu LY, Ma JX, Wang Y, Zhao J, Lu B, Ma XL. Adductor canal block versus continuous femoral nerve block in primary total knee arthroplasty: A meta-analysis. Int J Surg. 2016 Jul;31:17-24. doi: 10.1016/j.ijsu.2016.05.036. Epub 2016 May 19. PMID 27212592
- [Background] Grevstad U, Mathiesen O, Lind T, Dahl JB. Effect of adductor canal block on pain in patients with severe pain after total knee arthroplasty: a randomized study with individual patient analysis. Br J Anaesth. 2014 May;112(5):912-9. doi: 10.1093/bja/aet441. Epub 2014 Jan 8. PMID 24401802
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Background] Dong CC, Dong SL, He FC. Comparison of Adductor Canal Block and Femoral Nerve Block for Postoperative Pain in Total Knee Arthroplasty: A Systematic Review and Meta-analysis. Medicine (Baltimore). 2016 Mar;95(12):e2983. doi: 10.1097/MD.0000000000002983. PMID 27015172
- [Background] Hussain N, Ferreri TG, Prusick PJ, Banfield L, Long B, Prusick VR, Bhandari M. Adductor Canal Block Versus Femoral Canal Block for Total Knee Arthroplasty: A Meta-Analysis: What Does the Evidence Suggest? Reg Anesth Pain Med. 2016 May-Jun;41(3):314-20. doi: 10.1097/AAP.0000000000000376. No abstract available. PMID 27035459
- [Background] Li D, Yang Z, Xie X, Zhao J, Kang P. Adductor canal block provides better performance after total knee arthroplasty compared with femoral nerve block: a systematic review and meta-analysis. Int Orthop. 2016 May;40(5):925-33. doi: 10.1007/s00264-015-2998-x. Epub 2015 Oct 10. PMID 26452678
- [Background] Vora MU, Nicholas TA, Kassel CA, Grant SA. Adductor canal block for knee surgical procedures: review article. J Clin Anesth. 2016 Dec;35:295-303. doi: 10.1016/j.jclinane.2016.08.021. Epub 2016 Oct 11. PMID 27871547
- [Background] Ma J, Gao F, Sun W, Guo W, Li Z, Wang W. Combined adductor canal block with periarticular infiltration versus periarticular infiltration for analgesia after total knee arthroplasty. Medicine (Baltimore). 2016 Dec;95(52):e5701. doi: 10.1097/MD.0000000000005701. PMID 28033266